CLINICAL TRIAL: NCT03344328
Title: Evaluation of the Prevalence, Intensity and Consequences of Bortezomib-induced Neuropathic Disorders: Monocentric Observational and Cross-sectional Study.
Brief Title: Prevalence, Intensity and Consequences of Bortezomib-induced Neuropathic Disorders.
Acronym: PREVIB
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-359
Record Dates: First submitted 2017-10-18; First posted 2017-11-17 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2019-06

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy; Multiple Myeloma
Keywords: Chemotherapy; Bortezomib; Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Bortezomib — The algorithm (computer query) will identify all patients who received bortezomib-based chemotherapy for the multiple myeloma indication between 2008 and 2016. All the questionnaires used are validated in the scientific literature.

SUMMARY:
Cancer-induced peripheral neuropathies (CIPN) remain a real problem in oncology (Balayssac et al., 2011). These CIPN are induced by certain classes of anticancer drugs such as taxanes (paclitaxel and docetaxel), platinum salts (cisplatin and oxaliplatin), alkaloids of Madagascar periwinkle (vincristine), bortezomib, thalidomide and eribulin (Balayssac et al., 2011; Vahdat et al., 2013). These CIPN essentially translate into sensory disorders such as paresthesia, dysesthetics or numbness. More rarely, these CIPN may be associated with motor or vegetative disorders (Balayssac et al., 2011). According to the recent meta-analysis by Hershman et al., no treatment can be proposed as a "gold standard" for preventing or treating CIPN (Hershman et al., 2014). As a result, oncologists reduce or stop doses of neurotoxic anticancer drugs because patients with CIPN have a marked deterioration in quality of life and co-morbidities such as anxiety, depression and sleep disorders (Hong et al., 2014; Mols et al., 2014). Therefore, understanding the pathophysiology of CIPN is essential to propose new therapeutic strategies.

Among neurotoxic anticancer drugs, bortezomib remains relatively little studied in terms of pathophysiology compared to platinum salts or taxanes, while the neurotoxicity of bortezomib remains a limiting factor in treatment. Since 2012, the FDA and EMA have validated the administration of bortezomib subcutaneously instead of intravenously in order to limit the neurotoxicity of bortezomib (Minarik et al., 2015). Indeed, a large study (N=222) reported that subcutaneous administration of bortezomib allowed the same therapeutic efficacy to be maintained while improving the safety profile and in particular limiting peripheral neuropathies (CIPN all grades: 38% vs. 53%, p=0.044, grade> 2: 24% vs. 41%, p=0.012 and grade> 3: 6% vs. 16%, p=0.026) However, a recent retrospective study (N=446) reports that the prevalence of bortezomib-induced peripheral neuropathies after subcutaneous administration remains relatively high: all grade: 41%, grade> 2: 18%, grade> 3: 4%, and above all that this prevalence is not different between subcutaneous and intravenous routes (Minarik et al., 2015).

DETAILED DESCRIPTION:
Only 2 studies evaluated quantitatively and qualitatively the sensitivity disorders in patients with bortezomib-induced peripheral neuropathy by intravenous (Boyette-Davis et al., 2011; Cata et al., 2007). In these 2 studies, the patients presented a distribution of the sensitive disorders characteristic of the so-called stocking-glove distribution of the CIPN affecting the distal extremities of the limbs. A quantification of the sensory thresholds (QST) was carried out and revealed a number of sensitive anomalies. Neuropathic patients suffer from deficits in tactile sensitivity and disorders of thermal sensitivity. In Cata et al. study, patients showed hypersensitivity to painful cold (CIPN patients vs. healthy controls: 10.4±2°C vs. 3±1°C, p<0.05), hot perception deficit (CIPN patients vs. healthy controls: 40.2±1.4°C vs. 37±0.74°C, p<0.05) and a painful hot sensitivity deficit. However, the cold sensory disorders would be more inconstant, because in neuropathic patients suffering from bortezomib-induced peripheral neuropathy, another study by the same team found only warm tactile and thermal sensory anomalies, but did not reveal a cold perception anomaly (Boyette-Davis et al., 2011). Finally, a few rare cases of bortezomib-induced hearing impairment have been described in the literature (Chim and Wong, 2008; Engelhardt et al., 2005). This ototoxicity is thought to be linked to an alteration in the functioning of peroxisomes (Lee et al., 2015).

No studies have actually evaluated the long-term prevalence of bortezomib-induced neuropathy. The only studies with long-term follow-up have carried out a cumulative assessment over 22 months (Pantani et al., 2014), 32 months (Dimopoulos et al., 2013) and 60 months (Wang et al., 2016) of the therapeutic response and adverse reactions induced by bortezomib. No studies dedicated to neurological adverse events have been conducted in the long term. Thus, the prevalence, duration, intensity and reversibility of bortezomib-induced neuropathy are poorly known in the long term (more than 5 years). On the other hand, a measurement tool such as the QLQ-CIPN20 questionnaire (EORTC) evaluating the intensity of sensory, motor and vegetative disorders associated with CIPN, a questionnaire presented as the most specific tool in the evaluation of CIPN (Lavoie Smith et al., 2013; Postma et al., 2005), has never been tested in this patient population.

This study project aims to provide precise knowledge on the prevalence, intensity and consequences of bortezomib-induced neuropathy in the short (2016-2014) and medium (2014-2012) term after subcutaneous injection and in the long term (2012-2008) after intravenous injection, knowing that at the Clermont-Ferrand University Hospital, the route of administration of bortezomib was intravenous. Retreat to at least 9 years of age could provide information on the kinetics of onset and disappearance of neuropathy after chemotherapy treatments (data unknown in the literature to date). Finally, these data acquired in a French context relating to bortezomib-induced neuropathy may be used in future studies evaluating new intervention strategies to prevent and/or treat bortezomib-induced neuropathy.

This observational study will combine retrospective treatment data from the CHIMIO® chemotherapy prescribing software with data obtained from patients by answering questionnaires.

Patients will be identified from the CHIMIO® chemotherapy prescription software database. The algorithm (computer query) will identify all patients who received bortezomib-based chemotherapy for the multiple myeloma indication between 2008 and 2016. All the questionnaires used are validated in the scientific literature.

ELIGIBILITY:
Inclusion Criteria:

* - Patients previously treated with bortezomib for multiple myeloma between 2008 and 2016 at Clermont-Ferrand University Hospital.
* Oral non-opposition of participation in the study

Exclusion Criteria:

* Patient unable to understand or answer questionnaires.
* Age < 18 years.
* Neurological pathologies (e. g. Parkinson's syndrome, stroke, fibromyalgia, etc.).
* Legal incapacity (person deprived of liberty or under guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously treated with bortezomib for multiple myeloma between 2008 and 2016 at Clermont-Ferrand University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of peripheral neuropathy | at day 1
  Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20 (QLQ-CIPN20 ; EORTC- European Organisation for Research and Treatment of Cancer).
  The questionnaire is divided in 3 subscales: sensory, motor and vegetative. Severity scores summed from 0 to 100. A high score will correspond to the worst symptoms.
  * Sensory score CIPN20 ≤ 6 = grade 0 NCI-CTCAE
  * Sensory score CIPN20 > 6 and < 30 = grade 1 NCI-CTCAE
  * Sensory score CIPN20 ≥ 30 and < 80 = grade 2-3 NCI-CTCAE
  * Sensory score CIPN20 ≥ 80 = grade 4 NCI-CTCAE.

SECONDARY OUTCOMES:
Chronic pain | at day 1
  Pain score rated by a Visual Analog Scale (VAS, 0 (no pain) - 10 (worst possible pain)). Pain will be defined for a score of 4/10.
Screening of neuropathic pain | at day 1
  DN4 questionnaire interview (positive score> 3/7), if VAS pain> 4
Anxiety and Depression Score | at day 1
  Hospital Anxiety and Depression Scale (HADS, summed score from 0 to 21). Score ≤ 7 = no symptomatology, score between 8-10 = suspect symptomatology and score ≥ 11 = consistent symptomatology.
Hearing disorders | at day 1
  EVA and questions exploring possible hearing problems (professional or leisure activity exposing to noise, habit of having people repeat themselves, problems with telephone comprehension, need to increase television volume, difficulty following a conversation in the presence of noise).
Health -related quality of life related to chemotherapy treatment. | at day 1
  Quality of Life Questionnaire - Chemotherapy 30 (QLQ-C30, EORTC-European Organisation for Research and Treatment of Cancer).
  The questionnaire is divided in 3 subscales: Global health, functional and symptomatic.
  Severity scores summed from 0 to 100. For the global health scale and the functional scale, a high score will correspond to a better quality of life. For the symptomatic scale, a high score will correspond to a lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: David BALAYSSAC, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Giraudet F, Selvy M, Kerckhove N, Pereira B, Barreau F, Nguyen D, Busserolles J, Cabrespine A, Chaleteix C, Soubrier M, Bay JO, Lemal R, Balayssac D. Relation between auditory difficulties and bortezomib-induced peripheral neuropathy in multiple myeloma: a single-center cross-sectional study. Eur Arch Otorhinolaryngol. 2022 Apr;279(4):2197-2201. doi: 10.1007/s00405-021-07234-1. Epub 2022 Jan 31. PMID 35098333
- [Derived] Engelhardt M, Ihorst G, Singh M, Rieth A, Saba G, Pellan M, Lebioda A. Real-World Evaluation of Health-Related Quality of Life in Patients With Multiple Myeloma From Germany. Clin Lymphoma Myeloma Leuk. 2021 Feb;21(2):e160-e175. doi: 10.1016/j.clml.2020.10.002. Epub 2020 Oct 24. PMID 33218965